CLINICAL TRIAL: NCT07352631
Title: Efficacy and Safety of a Novel 532-nm Picosecond Nd:YAG Laser for the Treatment of Freckles in Chinese Patients: A Prospective, Randomized, Split-Face Controlled Study
Brief Title: A Novel 532-nm Picosecond Laser for Freckle Treatment in Chinese Patients
Acronym: PICO-FRECK-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MLDPMQB-01; MLDPMQB-01 (Registry Identifier: Nanjing Maidland Healthcare Co., Ltd)
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Freckles
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Laser Device (Experimental): Participants received treatment with the investigational Nd:YAG picosecond laser therapy device (Model: MLD picolander). The device emits light at a wavelength of 532 nm and was used according to the manufacturer's instructions and clinical judgment to treat freckles in the designated target area on one side of the face.
  Interventions: Device: Nd:YAG Picosecond Laser Therapy Device
- Control Laser Device (Active Comparator): Participants received treatment with the active control device, the marketed Nd:YAG picosecond laser therapy system (Model: PicoWay). This device also emits light at a wavelength of 532 nm and was used according to its approved instructions and clinical judgment to treat freckles in the symmetrical target area on the contralateral side of the face.
  Interventions: Device: Nd:YAG Picosecond Laser Therapy System

INTERVENTIONS:
Device: Nd:YAG Picosecond Laser Therapy Device — This is an investigational medical device. It is a Nd:YAG laser system that generates picosecond-duration pulses of light at a wavelength of 532 nanometers (nm). It is designed for the treatment of benign epidermal pigmented lesions, including freckles, through selective photothermolysis and photomechanical effects.
  Arms: Investigational Laser Device
Device: Nd:YAG Picosecond Laser Therapy System — This is a marketed (approved) medical device used as an active comparator. It is a Nd:YAG laser system that generates picosecond-duration pulses of light at a wavelength of 532 nanometers (nm). It is indicated for the treatment of benign epidermal pigmented lesions, including freckles.
  Arms: Control Laser Device

SUMMARY:
The goal of this clinical trial was to learn if a novel laser device works as well and is as safe as an already approved laser device for removing freckles on the face.

The main questions it aimed to answer were:

After 8 weeks, did the novel laser make freckles fade by 60% or more for a similar number of participants as the approved laser? What side effects did participants have from either laser? Researchers compared the results from two sides of each participant's face to see if the novel laser worked as well as the approved laser. One side of the face was treated with the novel laser, and the other side was treated with the approved laser. A computer randomly chose which side received which laser.

Participants in this study:

Were adults (aged 18-65) with similar freckles on both sides of their face. Received one laser treatment session, using the two different lasers on opposite sides of their face.

Returned to the clinic for check-up visits about 4 weeks and 8 weeks after the treatment.

Had photos taken of their face at each visit so doctors could compare the fading of their freckles.

Answered questions about any pain during the treatment and their satisfaction with the results.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years (inclusive).
* Fitzpatrick skin type III, IV, or V.
* Diagnosed with facial freckles.
* Presence of visually symmetrical bilateral facial freckles.
* Able to understand and voluntarily sign the informed consent form.
* Willing and able to comply with all study procedures and follow-up visits.

Exclusion Criteria:

* High photosensitivity to any light spectrum.
* Severe organic diseases (e.g., epilepsy, psychosis).
* History of sunburn within the past 1 month.
* History of skin malignancies (e.g., squamous cell carcinoma, melanoma).
* Skin lesions that are broken, inflamed, or with a history of poor wound healing or keloids.
* Diagnosis of cutaneous lupus erythematosus.
* Significant systemic disease or obvious lesions in the treatment area.
* Presence of herpes simplex virus (HSV) in the expected treatment area.
* Active local or systemic infection, or open wounds in the treatment area.
* History of immunosuppression/immunodeficiency (including HIV/AIDS) or use of immunosuppressive drugs.
* Use of anticoagulants or medications that may alter wound healing within the past 1 month.
* Use of known photosensitizing medications within the past 1 month.
* Oral isotretinoin (Accutane) use within 12 months prior to initial treatment or planned use during the study.
* Use of iron supplements, herbal supplements (e.g., Ginkgo, Ginseng, Garlic), or fish oil supplements within the past 1 month.
* Other photo or energy-based aesthetic procedures in the treatment area within the past 1 month.
* Pregnancy, lactation, or planning pregnancy during the study period.
* Participation in another clinical trial (except registry studies) within 3 months prior to screening.
* Considered by the investigator to have poor compliance or otherwise unsuitable for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Treatment Response Rate at 8 Weeks | 8 weeks after the single treatment session
  The proportion of participants achieving a treatment response at the 8-week follow-up visit. A response is defined as a lesion clearance rate of 60% or greater. The clearance rate is calculated as: [(Number of freckles at baseline - Number of freckles at 8 weeks) / Number of freckles at baseline] x 100%. Assessment is performed by blinded evaluators based on standardized photographs.

SECONDARY OUTCOMES:
Complete Clearance Rate at 8 Weeks | 8 weeks after the single treatment session
  The proportion of participants achieving complete clearance of freckles at the 8-week follow-up visit. Complete clearance is defined as a lesion clearance rate of 90% or greater. The clearance rate is calculated as: [(Number of freckles at baseline - Number of freckles at 8 weeks) / Number of freckles at baseline] x 100%. Assessment is performed by blinded evaluators based on standardized photographs.
Global Aesthetic Improvement Scale (GAIS) Score at 8 Weeks | 8 weeks after the single treatment session
  The overall improvement in aesthetic appearance of the treated areas as assessed by blinded evaluators at the 8-week follow-up visit, using the Global Aesthetic Improvement Scale (GAIS). The GAIS is a 5-point scale ranging from 1 (Worse) to 5 (Very Much Improved).
Pain Score During Treatment (VAS) | Immediately after the single treatment session (within 30 minutes)
  The level of pain experienced by participants during the laser treatment, assessed immediately (within 30 minutes) after the treatment using a Visual Analogue Scale (VAS). The VAS is a continuous scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Participant Satisfaction Score at 8 Weeks | 8 weeks after the single treatment session
  The degree of participant satisfaction with the treatment results regarding pigment clearance, assessed at the 8-week follow-up visit using a satisfaction survey. The score ranges from 1 (completely dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Bengbu First People's Hospital, Bengbu, Anhui
  - Beijing Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
1. Privacy and Confidentiality: The data contain sensitive personal health information of participants, and sharing such data may compromise participant privacy and confidentiality.
  2. Commercial and Regulatory Constraints: The trial is sponsored by a medical device company, and the data are subject to intellectual property protection and ongoing regulatory review processes.
  3. Lack of Data Sharing Mechanism: There is currently no established infrastructure or agreement for external data sharing in this trial.

REFERENCES:
- See also: Related Info — http://www.bioray-med.com